CLINICAL TRIAL: NCT02329730
Title: Phase IIa Clinical Study of Recombinant Mycobacterium Tuberculosis Antigen ESAT6-CFP10
Brief Title: Phase IIa Clinical Study of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Shanghai Public Health Clinical Center (Other Government); Tianjin Haihe Hospital (Other); Air Force Military Medical University, China (Other); Proswell Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LTao-EC IIa
Record Dates: First submitted 2014-12-23; First posted 2015-01-01 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-03

CONDITIONS: Tuberculosis
Keywords: diagnosis of Tuberculosis (TB); ESAT6; CFP10; Phase IIa Clinical Trial
MeSH Terms: conditions — Tuberculosis | interventions — Tuberculin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- the healthy subjects (Experimental): The healthy subjects inject 1μg/ml ESAT6-CFP10 and tuberculin purified protein derivative only one time , or 5μg/ml ESAT6-CFP10 and tuberculin purified protein derivative only one time , or 10μg/ml ESAT6-CFP10 and tuberculin purified protein derivative only one time , or 20μg/ml ESAT6-CFP10 and tuberculin purified protein derivative only one time .Right arm inject ESAT6-CFP10 and left arm inject tuberculin purified protein derivative. Two drugs must be use in the same subjects.
  Interventions: Biological: 1μg/ml ESAT6-CFP10 and tuberculin purified protein derivative; Biological: 5μg/ml ESAT6-CFP10 and tuberculin purified protein derivative; Biological: 10μg/ml ESAT6-CFP10 and tuberculin purified protein derivative; Biological: 20μg/ml ESAT6-CFP10 and tuberculin purified protein derivative
- the first part of tuberculosis subjects (Experimental): The first part kind of tuberculosis subjects inject 1μg/ml ESAT6-CFP10 and tuberculin purified protein derivative only one time , or 5μg/ml ESAT6-CFP10 and tuberculin purified protein derivative only one time , or 10μg/ml ESAT6-CFP10 and tuberculin purified protein derivative only one time , or 20μg/ml ESAT6-CFP10 and tuberculin purified protein derivative only one time .Right arm inject ESAT6-CFP10 and left arm inject tuberculin purified protein derivative. Two drugs must be use in the same subjects.
  Interventions: Biological: 1μg/ml ESAT6-CFP10 and tuberculin purified protein derivative; Biological: 5μg/ml ESAT6-CFP10 and tuberculin purified protein derivative; Biological: 10μg/ml ESAT6-CFP10 and tuberculin purified protein derivative; Biological: 20μg/ml ESAT6-CFP10 and tuberculin purified protein derivative
- the second part of tuberculosis subjects (Experimental): The second part of tuberculosis subjects inject 1μg/ml ESAT6-CFP10 and placebo only one time , or 5μg/ml ESAT6-CFP10 and placebo only one time , or 10μg/ml ESAT6-CFP10 and placebo only one time , or 20μg/ml ESAT6-CFP10 and placebo only one time .Right arm inject ESAT6-CFP10 and left arm inject placebo. Two drugs must be use in the same subjects.
  Interventions: Biological: 1μg/ml ESAT6-CFP10 and placebo; Biological: 5μg/ml ESAT6-CFP10 and placebo; Biological: 10μg/ml ESAT6-CFP10 and placebo; Biological: 20μg/ml ESAT6-CFP10 and placebo

INTERVENTIONS:
Biological: 1μg/ml ESAT6-CFP10 and tuberculin purified protein derivative — Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal injection 1μg/ml ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 Allergen and TB-PPD only one time in the healthy subjects and the first part of tuberculosis subjects respectively.
  Other Names: Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 /TB-PPD
  Arms: the first part of tuberculosis subjects; the healthy subjects
Biological: 5μg/ml ESAT6-CFP10 and tuberculin purified protein derivative — Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal injection 5g/ml ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 Allergen and TB-PPD only one time in the healthy subjects and the first part of tuberculosis subjects respectively.
  Other Names: Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10/TB-PPD
  Arms: the first part of tuberculosis subjects; the healthy subjects
Biological: 10μg/ml ESAT6-CFP10 and tuberculin purified protein derivative — Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal injection 10g/ml ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 Allergen and TB-PPD only one time in the healthy subjects and the first part of tuberculosis subjects respectively.
  Other Names: Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 /TB-PPD
  Arms: the first part of tuberculosis subjects; the healthy subjects
Biological: 20μg/ml ESAT6-CFP10 and tuberculin purified protein derivative — Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal injection 20/ml ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 Allergen and TB-PPD only one time in the healthy subjects and the first part of tuberculosis subjects respectively.
  Other Names: Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 /TB-PPD
  Arms: the first part of tuberculosis subjects; the healthy subjects
Biological: 1μg/ml ESAT6-CFP10 and placebo — Left arm intradermal injection of the placebo of 1μg/ml ESAT6-CFP10 by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal injection 1μg/ml ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 and placebo only one time in the second part of tuberculosis subjects.
  Other Names: Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10
  Arms: the second part of tuberculosis subjects
Biological: 5μg/ml ESAT6-CFP10 and placebo — Left arm intradermal injection of the placebo of 5μg/ml ESAT6-CFP10 by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal injection 5μg/ml ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 and placebo only one time in the second part of tuberculosis subjects.
  Other Names: Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10
  Arms: the second part of tuberculosis subjects
Biological: 10μg/ml ESAT6-CFP10 and placebo — Left arm intradermal injection of the placebo of 10μg/ml ESAT6-CFP10 by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal injection 10μg/ml ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 and placebo only one time in the second part of tuberculosis subjects.
  Other Names: Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10
  Arms: the second part of tuberculosis subjects
Biological: 20μg/ml ESAT6-CFP10 and placebo — Left arm intradermal injection of the placebo of 20μg/ml ESAT6-CFP10 by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal injection 20μg/ml ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 and placebo only one time in the second part of tuberculosis subjects.
  Other Names: Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10
  Arms: the second part of tuberculosis subjects

SUMMARY:
Choose healthy subjects and patients with TB, distribute them into different dose groups according to the recombinant EC allergen dose from low to high average. Conducting clinical trials of TB-PPD or placebo as controlled arms intradermal injection. Do specific interferon gamma detection before the skin test，after the test 72h±2h and 144h±2h. Evaluate the safety of the recombinant EC allergy , and provide the appropriate dose range for phase IIb clinical trials.

DETAILED DESCRIPTION:
First, 56 healthy subjects are distributed into different dose groups according to the recombinant EC allergen dose from low to high.Conducting clinical trials of TB-PPD as controlled arms intradermal injection.Do specific interferon gamma detection before the skin test，after the test 72h±2h and 144h±2h. The vital signs (breathing, heart rate, blood pressure and temperature), skin reaction at injection site (flush and induration) , local reactions (rash, pain, itching and skin mucous membrane) and a variety of adverse events; The vital signs, blood routine, urine routine, liver and kidney function, electrocardiogram （before the skin test,after skin test 144h ）are the main test items,Evaluate the safety of the recombinant EC allergy in the expansion of the healthy people , and provide the appropriate dose range for phase IIb clinical trials.

Second，56 patients of TB are distributed different dose groups according to the recombinant EC allergen dose from low to high. Conducting clinical trials of TB-PPD as controlled arms intradermal injection.Do specific interferon gamma detection before the skin test，after the test 72h±2h and 144h±2h. The vital signs (breathing, heart rate, blood pressure and temperature),skin reaction at injection site (flush and induration) , local reactions (rash, pain, itching and skin mucous membrane) and a variety of adverse events; The vital signs, blood routine, urine routine, liver and kidney function, electrocardiogram （before the skin test,after skin test 144h ）are the main test items,Evaluate the safety of the recombinant EC allergy in patients of TB,and provide the appropriate dose range for phase IIb clinical trials.

Third，32 patients of TB are distributed into different dose groups according to the recombinant EC allergen dose from low to high. Conducting clinical trials of placebo as controlled arms intradermal injection.Do specific interferon gamma detection before the skin test，after the test 72h±2h and 144h±2h. The vital signs (breathing, heart rate, blood pressure and temperature), skin reaction at injection site (flush and induration), local reactions (rash, pain, itching and skin mucous membrane) and a variety of adverse events; The vital signs, blood routine, urine routine, liver and kidney function, electrocardiogram （before the skin test,after skin test 144h ）are the main test items,Evaluate the safety of the recombinant EC allergy in patients of TB on safety.

ELIGIBILITY:
Inclusion Criteria of healthy subjects:

1. 18 to 65 years old
2. Consent and signed ICF(informed consent forms)
3. Comply with follow-up
4. No history or family history of TB(tuberculosis)
5. Without the internal and external of pulmonary tuberculosis ; no symptoms of respiratory tract and other body parts for TB
6. The examination such as X-ray chest radiograph, sputum bacteria confirmed non-tuberculosis (TB)
7. No uncontrolled kinds of acute or chronic disease or acute infectious diseases or skin disease or skin allergies due to a variety of causes
8. Physical condition : No obvious heart, liver, kidney, gastrointestinal tract, nervous system, mental disorder and metabolic abnormalities and other medical history from signed informed consent to the injection within four weeks prior to delivery ;by the comprehensive physical examination showed electrocardiogram, blood pressure, heart rate, breathing and laboratory tests, including blood, urine routine, liver, kidney and other various biochemical test all without exception or slightly unusual but does not affect our research
9. Did not attend any other new drug clinical trials and not vaccinate prevention products and immunoglobulin for nearly 3 months
10. Normal axillary temperature(quiet condition ≤37.0 ℃)
11. No smoking, no alcohol and drinking caffeinated beverages during the study

Exclusion Criteria of Healthy volunteers:

1. Has the following serious disease, such as advanced cancer, diabetes, chronic obstructive pulmonary disease (copd) in acute episodes, acute/ progressive liver disease or kidney disease, congestive heart failure, etc
2. Have seizures, epilepsy, brain and nervous system symptoms or signs of history
3. Has known or suspected (or risk possible) immune damaged or abnormal functional , accept glucocorticoid and immunosuppressants or immunopotentiator treatment, outside the gastrointestinal tract protein or blood products or plasma extraction in 3 months, immunodeficiency virus infection or related diseases
4. Has acute febrile diseases and infectious diseases
5. Participate in other new drug clinical trials
6. Participated in any other new drug clinical trials in 3 months
7. Allergic people who have histories of allergy to two or more drugs/food allergy and physical scars, are allergic to alcohol or drugs known to the group of points
8. Women who are in pregnancy or lactation
9. People with mental or physical disabilities
10. Researchers consider that any conditions may affect the trial evaluation

Inclusion Criteria of TB (tuberculosis)subjects:

1. Diagnosis TB according to the health of the People's Republic of China industry standard WS 288-2008 tuberculosis diagnostic criteria
2. Aged 18 to 65 years old
3. Consent and signed ICF to participate in this study
4. Comply with the requirements of the clinical research plan for follow-up

Exclusion Criteria of TB volunteers:

1. Have the following serious disease, such as advanced cancer, diabetes, chronic obstructive pulmonary disease (copd) in acute episodes, acute/ progressive liver disease or kidney disease, congestive heart failure, etc
2. Have seizures, epilepsy, brain and nervous system symptoms or signs of history;
3. Have known or suspected (or risk possible) immune damaged or abnormal functional , accept glucocorticoid and immunosuppressants or immunopotentiator treatment, outside the gastrointestinal tract protein or blood products or plasma extraction in 3 months, immunodeficiency virus infection or related diseases
4. People in the pyrogenic stage with febrile diseases or infectious diseases (non tuberculosis)
5. Participate in other new drug clinical trials
6. Participated in any other new drug clinical trials in 3 months;
7. Allergic people who have histories of allergy to two or more drugs/food allergy and physical scars, are allergic to alcohol or drugs known to the group of points;
8. Women who are in pregnancy or lactation;
9. People with mental or physical disabilities;
10. Researchers consider that any conditions may affect the trial evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuihua Lu, Bachelor, Principal Investigator — Shanghai Public Health Clinical Center; Qi Wu, Master, Principal Investigator — Tianjin Haihe Hospital

REFERENCES:
- [Background] van Pinxteren LA, Ravn P, Agger EM, Pollock J, Andersen P. Diagnosis of tuberculosis based on the two specific antigens ESAT-6 and CFP10. Clin Diagn Lab Immunol. 2000 Mar;7(2):155-60. doi: 10.1128/CDLI.7.2.155-160.2000. PMID 10702486
- [Background] Ravn P, Munk ME, Andersen AB, Lundgren B, Lundgren JD, Nielsen LN, Kok-Jensen A, Andersen P, Weldingh K. Prospective evaluation of a whole-blood test using Mycobacterium tuberculosis-specific antigens ESAT-6 and CFP-10 for diagnosis of active tuberculosis. Clin Diagn Lab Immunol. 2005 Apr;12(4):491-6. doi: 10.1128/CDLI.12.4.491-496.2005. PMID 15817755
- [Background] Brusasca PN, Colangeli R, Lyashchenko KP, Zhao X, Vogelstein M, Spencer JS, McMurray DN, Gennaro ML. Immunological characterization of antigens encoded by the RD1 region of the Mycobacterium tuberculosis genome. Scand J Immunol. 2001 Nov;54(5):448-52. doi: 10.1046/j.1365-3083.2001.00975.x. PMID 11696195
- [Background] Weldingh K, Andersen P. ESAT-6/CFP10 skin test predicts disease in M. tuberculosis-infected guinea pigs. PLoS One. 2008 Apr 23;3(4):e1978. doi: 10.1371/journal.pone.0001978. PMID 18431468
- [Background] Aagaard C, Govaerts M, Meikle V, Vallecillo AJ, Gutierrez-Pabello JA, Suarez-Guemes F, McNair J, Cataldi A, Espitia C, Andersen P, Pollock JM. Optimizing antigen cocktails for detection of Mycobacterium bovis in herds with different prevalences of bovine tuberculosis: ESAT6-CFP10 mixture shows optimal sensitivity and specificity. J Clin Microbiol. 2006 Dec;44(12):4326-35. doi: 10.1128/JCM.01184-06. Epub 2006 Sep 27. PMID 17005738
- See also: Center for drug evaluation, CFDA ,China — https://wbca.cde.org.cn/wbca/clinmain.do?method=edit&ckmIdCode=8BE5738082A97A9E5471F80B4F814FCF

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Subjects-1μg/ml ESAT6-CFP10 & TB-PPD: The same healthy subjects inject 1μg/ml ESAT6-CFP10 and TB-PPD only one time .Right arm inject ESAT6-CFP10 and left arm TB-PPD.Two drugs must be use in the same subjects.
  Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 and TB-PPD only one time in every healthy subjects .
- Healthy Subjects-5μg/ml ESAT6-CFP10 & TB-PPD: The same healthy subjects inject 5μg/ml ESAT6-CFP10 and TB-PPD only one time .Right arm inject ESAT6-CFP10 and left arm TB-PPD.Two drugs must be use in the same subjects.
  Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject respectively ESAT6-CFP10 and TB-PPD only one time in every healthy subjects .
- Healthy Subjects-10μg/ml ESAT6-CFP10 & TB-PPD: The same healthy subjects inject 10μg/ml ESAT6-CFP10 and TB-PPD only one time .Right arm inject ESAT6-CFP10 and left arm TB-PPD.Two drugs must be use in the same subjects.
  Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject respectively ESAT6-CFP10 and TB-PPD only one time in every healthy subjects .
- Healthy Subjects-20μg/ml ESAT6-CFP10 & TB-PPD: The same healthy subjects inject 20μg/ml ESAT6-CFP10 and TB-PPD only one time .Right arm inject ESAT6-CFP10 and left arm TB-PPD.Two drugs must be use in the same subjects.
  Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject respectively ESAT6-CFP10 and TB-PPD only one time in every healthy subjects .
- Tuberculosis Subjects-1μg/ml ESAT6-CFP10 & TB-PPD: The same tuberculosis subjects inject 1μg/ml ESAT6-CFP10 and TB-PPD only one time .Right arm inject ESAT6-CFP10 and left arm TB-PPD.Two drugs must be use in the same subjects.
  Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject respectively ESAT6-CFP10 and TB-PPD only one time in every subjects .
- Tuberculosis Subjects-5μg/ml ESAT6-CFP10 & TB-PPD: The same tuberculosis subjects inject 5μg/ml ESAT6-CFP10 and TB-PPD only one time .Right arm inject ESAT6-CFP10 and left arm TB-PPD.Two drugs must be use in the same subjects.
  Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject respectively ESAT6-CFP10 and TB-PPD only one time in every subjects .
- Tuberculosis Subjects-10μg/ml ESAT6-CFP10 & TB-PPD: The same tuberculosis subjects inject 10μg/ml ESAT6-CFP10 and TB-PPD only one time .Right arm inject ESAT6-CFP10 and left arm TB-PPD.Two drugs must be use in the same subjects.
  Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject respectively ESAT6-CFP10 and TB-PPD only one time in every subjects .
- Tuberculosis Subjects-20μg/ml ESAT6-CFP10 & TB-PPD: The same tuberculosis subjects inject 20μg/ml ESAT6-CFP10 and TB-PPD only one time .Right arm inject ESAT6-CFP10 and left arm TB-PPD.Two drugs must be use in the same subjects.
  Left arm intradermal injection of 0.1ml TB-PPD(50IU/ml) by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject respectively ESAT6-CFP10 and TB-PPD only one time in every subjects .
- Tuberculosis Subjects-1μg/ml ESAT6-CFP10 & Placebo: The tuberculosis subjects inject 1μg/ml ESAT6-CFP10 and placebo of ESAT6-CFP10 only one time .Right arm inject ESAT6-CFP10 and left arm inject placebo. Two drugs must be use in the same subjects.
  Left arm intradermal injection of the placebo of ESAT6-CFP10 by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 and placebo only one time in same tuberculosis subjects.
- Tuberculosis Subjects-5μg/ml ESAT6-CFP10 & Placebo: The tuberculosis subjects inject 5μg/ml ESAT6-CFP10 and placebo of ESAT6-CFP10 only one time .Right arm inject ESAT6-CFP10 and left arm inject placebo. Two drugs must be use in the same subjects.
  Left arm intradermal injection of the placebo of ESAT6-CFP10 by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 and placebo only one time in same tuberculosis subjects.
- Tuberculosis Subjects-10μg/ml ESAT6-CFP10 & Placebo: The tuberculosis subjects inject 10μg/ml ESAT6-CFP10 and placebo of ESAT6-CFP10 only one time .Right arm inject ESAT6-CFP10 and left arm inject placebo. Two drugs must be use in the same subjects.
  Left arm intradermal injection of the placebo of ESAT6-CFP10 by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 and placebo only one time in same tuberculosis subjects.
- Tuberculosis Subjects-20μg/ml ESAT6-CFP10 & Placebo: The tuberculosis subjects inject 20μg/ml ESAT6-CFP10 and placebo of ESAT6-CFP10 only one time .Right arm inject ESAT6-CFP10 and left arm inject placebo. Two drugs must be use in the same subjects.
  Left arm intradermal injection of the placebo of ESAT6-CFP10 by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermal inject ESAT6-CFP10 by a syringe(1ml). Inject ESAT6-CFP10 and placebo only one time in same tuberculosis subjects.
Period: Overall Study
Arm/Group | Healthy Subjects-1μg/ml ESAT6-CFP10 & TB-PPD | Healthy Subjects-5μg/ml ESAT6-CFP10 & TB-PPD | Healthy Subjects-10μg/ml ESAT6-CFP10 & TB-PPD | Healthy Subjects-20μg/ml ESAT6-CFP10 & TB-PPD | Tuberculosis Subjects-1μg/ml ESAT6-CFP10 & TB-PPD | Tuberculosis Subjects-5μg/ml ESAT6-CFP10 & TB-PPD | Tuberculosis Subjects-10μg/ml ESAT6-CFP10 & TB-PPD | Tuberculosis Subjects-20μg/ml ESAT6-CFP10 & TB-PPD | Tuberculosis Subjects-1μg/ml ESAT6-CFP10 & Placebo | Tuberculosis Subjects-5μg/ml ESAT6-CFP10 & Placebo | Tuberculosis Subjects-10μg/ml ESAT6-CFP10 & Placebo | Tuberculosis Subjects-20μg/ml ESAT6-CFP10 & Placebo
Started | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 8 | 8 | 8 | 8
Completed | 14 | 14 | 14 | 14 | 11 | 12 | 13 | 13 | 7 | 7 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Each group of baseline analysis population apply full analysis set (FAS).FAS are the participant, following the principle of ITT, who receive at least once drug and have curative effect evaluation of drug treatment .Missing data of the curative effect part in FAS population use Last observation carried forward(LOCF)method to supplement.
Groups:
- 1μg/ml ESAT6-CFP10: The healthy subjects and TB subjects inject 1μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) or the placebo of ESAT6-CFP10 only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD or the placebo .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml) or the placebo by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 or the placebo of ESAT6-CFP10 by a syringe(1ml).
- 5μg/ml ESAT6-CFP10: The healthy subjects and TB subjects inject 5μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) or the placebo of ESAT6-CFP10 only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD or the placebo .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml) or the placebo by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 or the placebo of ESAT6-CFP10 by a syringe(1ml).
- 10μg/ml ESAT6-CFP10: The healthy subjects and TB subjects inject 10μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) or the placebo of ESAT6-CFP10 only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD or the placebo .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml) or the placebo by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 or the placebo of ESAT6-CFP10 by a syringe(1ml).
- 20μg/ml ESAT6-CFP10: The healthy subjects and TB subjects inject 20μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) or the placebo of ESAT6-CFP10 only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD or the placebo .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml) or the placebo by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 or the placebo of ESAT6-CFP10 by a syringe(1ml).
- Total: Total of all reporting groups
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10 | Total
Number analyzed (Participants) | 35 | 34 | 36 | 36 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.12 (12.83) | 38.46 (11.98) | 43.81 (12.53) | 44.63 (12.37) | 41.76 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 16 | 17 | 70
  Male | 18 | 14 | 20 | 19 | 71
height [Mean (Standard Deviation); unit: cm] | 166.83 (7.06) | 166.32 (7.59) | 167.44 (8.23) | 165.47 (7.81) | 166.52 (7.67)
weight [Mean (Standard Deviation); unit: kg] | 62.20 (9.70) | 62.15 (9.83) | 59.33 (9.40) | 59.42 (11.56) | 60.78 (10.12)

OUTCOME MEASURES:

1. Primary Outcome: Number of Healthy Participants Negative for Reaction at 24 Hours After Intradermal Injection With ESAT6-CFP10
Description: The investigators measure the longitudinal diameter and transverse diameter of induration and/or redness of ESAT6-CFP10 in healthy participants at 24 hours after intradermal injection by vernier caliper . And at the same blisters and lymphangitis are the specificity of the positive reaction of ESAT6-CFP10 .So induration ,redness ,blisters and lymphangitis in the healthy participants' arm are positive reaction.
  The percentage of negative(negative number/total number*100%) is the specificity of ESAT6-CFP10 .
Time Frame: 24 hours after intradermal injection
Population: The percentage of negative(negative number/total number*100%) is the specificity of ESAT6-CFP10 .
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 14 | 14 | 14 | 14
participants | 13 | 13 | 14 | 13

2. Secondary Outcome: the Number of Participants With Adverse Events
Description: evaluate specific time point of vital signs, skin test reaction, blood routine, urine routine, liver and kidney function, electrocardiogram and adverse events as the incidence of adverse events in the participants .
  Skin test reaction observation time: at the end of the skin test, skin test after 15 minutes, 1 hour, 4 hours, 24 hours, 48 hours, 72 hours, 96 hours; Vital signs evaluation time: 0 minutes before the subjects were intradermal injection, intradermal injection after 15 minutes, 1 hour, 4 hours, 24 hours, 48 hours, 72 hours, 96 hours, 144 hours.
  Blood routine, urine routine, liver and kidney function, electrocardiogram (ecg) evaluation time: skin test before and 144 h after injection; adverse events evaluation time: participants signed a written informed consent to finish all the follow-up.
Time Frame: before injection to 144 hours (plus or minus 2 hours) after injection
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 36 | 36 | 36 | 36
participants | 16 | 19 | 19 | 14

3. Secondary Outcome: the Number of Healthy Participants Negative for IFN-γ(Gamma Interferon ) Before Injection
Description: The investigator draw 5ml venous blood for detection of IFN-γ four hours before injection with drug.The percentage of negative(negative number/total number*100%) is the specificity of IFN-γ in healthy participants.
Time Frame: before injection and after signed ICF(informed consent forms)
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 14 | 14 | 14 | 14
participants | 12 | 13 | 13 | 13

4. Secondary Outcome: the Number of Tuberculosis (TB) Participants Positive for IFN-γ(Gamma Interferon ) Before Injection
Description: The investigator draw 5ml venous blood for detection of IFN-γ four hours before injection with drug. The percentage of positive(positive number/total number*100%) is the sensitivity of IFN-γ in TB Participants.
Time Frame: 4 hours before injection and after signed ICF(informed consent forms)
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 18 | 19 | 21 | 21
participants | 18 | 17 | 18 | 19

5. Secondary Outcome: the Number of Healthy Participants Negative for IFN-γ(Gamma Interferon ) at 72 Hours After Intradermal Injection With ESAT6-CFP10
Description: as for outcome 3
Time Frame: 72 hours after injection
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 14 | 14 | 14 | 14
participants | 13 | 12 | 13 | 13

6. Secondary Outcome: the Number of Tuberculosis (TB) Participants Positive for IFN-γ(Gamma Interferon ) at 72 Hours After Intradermal Injection With ESAT6-CFP10
Description: The investigator draw 5ml venous blood for detection of IFN-γ 72 hours after injection with drug.The percentage of positive(positivenumber/total number*100%) is the sensitivity of IFN-γ in in TB participants.
Time Frame: 72 hours after injection
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 18 | 19 | 21 | 21
participants | 18 | 19 | 18 | 19

7. Secondary Outcome: the Number of Healthy Participants Negative for IFN-γ(Gamma Interferon ) at 144 Hours After Intradermal Injection With ESAT6-CFP10
Description: The investigator draw 5ml venous blood for detection of IFN-γ 144 hours after injection with drug.The percentage of negative(negative number/total number*100%) is the specificity of IFN-γ in healthy participants.
Time Frame: 144 hours after injection
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 14 | 14 | 14 | 14
participants | 12 | 11 | 12 | 13

8. Secondary Outcome: the Number of Tuberculosis (TB) Participants Positive for IFN-γ(Gamma Interferon ) at 144 Hours After Intradermal Injection With ESAT6-CFP10
Description: The investigator draw 5ml venous blood for detection of IFN-γ 144 hours before injection with drug.The percentage of positive(positive number/total number*100%) is the sensitivity of IFN-γ in in TB participants.
Time Frame: 144 hours after injection
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 18 | 19 | 19 | 21
participants | 17 | 19 | 15 | 19

9. Primary Outcome: Number of Tuberculosis (TB) Participants Positive for Reaction at 24 Hours After Intradermal Injection With ESAT6-CFP10
Description: The investigators measure the longitudinal diameter and transverse diameter of induration and/or redness of ESAT6-CFP10 in TB participants at 24 hours after intradermal injection by vernier caliper . And at the same blisters and lymphangitis are the specificity of the positive reaction of ESAT6-CFP10 .So induration ,redness ,blisters and lymphangitis in the participants' arm are positive reaction.
Time Frame: 24 hours after intradermal injection
Population: The percentage of positive(positive number/total number*100%) is the sensitivity of ESAT6-CFP10 .
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 18 | 19 | 21 | 21
participants | 15 | 19 | 17 | 19

10. Primary Outcome: Number of Healthy Participants Negative for Reaction at 48 Hours After Intradermal Injection With ESAT6-CFP10
Description: The investigators measure the longitudinal diameter and transverse diameter of induration and/or redness of ESAT6-CFP10 in healthy participants at 48 hours after intradermal injection by vernier caliper . And at the same blisters and lymphangitis are the specificity of the positive reaction of ESAT6-CFP10 .So induration ,redness ,blisters and lymphangitis in the healthy participants' arm are positive reaction.
Time Frame: 48 hours after intradermal injection
Population: The percentage of negative(negative number/total number*100%) is the specificity of ESAT6-CFP10 .
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 14 | 14 | 14 | 14
participants | 13 | 13 | 13 | 13

11. Primary Outcome: Number of Tuberculosis (TB) Participants Positive for Reaction at 48 Hours After Intradermal Injection With ESAT6-CFP10
Description: The investigators measure the longitudinal diameter and transverse diameter of induration and/or redness of ESAT6-CFP10 in TB participants at 48 hours after intradermal injection by vernier caliper . And at the same blisters and lymphangitis are the specificity of the positive reaction of ESAT6-CFP10 .So induration ,redness ,blisters and lymphangitis in the participants' arm are positive reaction.
Time Frame: 48 hours after intradermal injection
Population: The percentage of positive(positive number/total number*100%) is the sensitivity of ESAT6-CFP10.
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 18 | 19 | 21 | 21
participants | 15 | 17 | 17 | 16

12. Primary Outcome: Number of Healthy Participants Negative for Reaction at 72 Hours After Intradermal Injection With ESAT6-CFP10
Description: The investigators measure the longitudinal diameter and transverse diameter of induration and/or redness of ESAT6-CFP10 in healthy participants at 72 hours after intradermal injection by vernier caliper . And at the same blisters and lymphangitis are the specificity of the positive reaction of ESAT6-CFP10 .So induration ,redness ,blisters and lymphangitis in the healthy participants' arm are positive reaction.
  The percentage of negative(negative number/total number*100%) is the specificity of ESAT6-CFP10
Time Frame: 72 hours after intradermal injection
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 14 | 14 | 14 | 14
participants | 13 | 13 | 13 | 13

13. Primary Outcome: Number of Tuberculosis (TB) Participants Positive for Reaction at 72 Hours After Intradermal Injection With ESAT6-CFP10
Description: The investigators measure the longitudinal diameter and transverse diameter of induration and/or redness of ESAT6-CFP10 in TB participants at 72 hours after intradermal injection by vernier caliper . And at the same blisters and lymphangitis are the specificity of the positive reaction of ESAT6-CFP10 .So induration ,redness ,blisters and lymphangitis in the participants' arm are positive reaction.
Time Frame: 72 hours after intradermal injection
Population: The percentage of positive(positive number/total number*100%) is the sensitivity of ESAT6-CFP10 .
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 18 | 19 | 21 | 21
participants | 15 | 17 | 17 | 16

14. Primary Outcome: Number of Healthy Participants Negative for Reaction at 96 Hours After Intradermal Injection With ESAT6-CFP10
Description: The investigators measure the longitudinal diameter and transverse diameter of induration and/or redness of ESAT6-CFP10 in healthy participants at 96 hours after intradermal injection by vernier caliper . And at the same blisters and lymphangitis are the specificity of the positive reaction of ESAT6-CFP10 .So induration ,redness ,blisters and lymphangitis in the healthy participants' arm are positive reaction.
Time Frame: 96 hours after intradermal injection
Population: The percentage of negative(negative number/total number*100%) is the specificity of ESAT6-CFP10 .
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 14 | 14 | 14 | 14
participants | 13 | 13 | 13 | 13

15. Primary Outcome: Number of Tuberculosis (TB) Participants Positive for Reaction at 96 Hours After Intradermal Injection With ESAT6-CFP10
Description: The investigators measure the longitudinal diameter and transverse diameter of induration and/or redness of ESAT6-CFP10 in TB participants at 96 hours after intradermal injection by vernier caliper . And at the same blisters and lymphangitis are the specificity of the positive reaction of ESAT6-CFP10 .So induration ,redness ,blisters and lymphangitis in the participants' arm are positive reaction.
Time Frame: 96 hours after intradermal injection
Population: The percentage of positive(positive number/total number*100%) is the sensitivity of ESAT6-CFP10 .
Measure: Number; unit: participants
Arm/Group | 1μg/ml ESAT6-CFP10 | 5μg/ml ESAT6-CFP10 | 10μg/ml ESAT6-CFP10 | 20μg/ml ESAT6-CFP10
Number analyzed (Participants) | 18 | 19 | 21 | 21
participants | 14 | 17 | 17 | 15

ADVERSE EVENTS:
Time Frame: We collect all kinds of adverse events related to the study drugs from signed ICF to the seventh day after injection with skin drugs.
Description: Every subjects inject two drug in the different time.Because the two drugs only interval 30 minutes ,adverse events related to the study drugs contain ESAT6-CFP10 ,placebo or TB-PPD in one participant.Related to study drug is refers to the relationship with the study drug "for sure about、 is likely to be relevant、 may be related to"。
Groups:
- Healthy Subjects-1μg/ml ECand TB-PPD: The healthy subjects inject 1μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml)by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
- Healthy Subjects-5μg/ml EC and TB-PPD: The healthy subjects inject 5μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml)by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
- Healthy Subjects-10μg/ml EC and TB-PPD: The healthy subjects inject 10μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml)by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
- Healthy Subjects-20μg/ml EC and TB-PPD: The healthy subjects inject 20μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml)by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
- Tuberculosis Subjects- 1μg/mlEC and TB-PPD: The tuberculosis subjects inject 1μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml)by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
- Tuberculosis Subjects- 5μg/ml EC and TB-PPD: The tuberculosis subjects inject 5μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml)by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
- Tuberculosis Subjects- 10μg/ml EC and TB-PPD: The tuberculosis subjects inject 10μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml)by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
- Tuberculosis Subjects- 20μg/ml EC and TB-PPD: The tuberculosis subjects inject 20μg/ml ESAT6-CFP10 and tuberculin purified protein derivative (TB-PPD) only one time in the different time .Right arm inject ESAT6-CFP10 and left arm inject TB-PPD .Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml TB-PPD(50IU/ml)by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
- Tuberculosis Subjects- 1μg/ml EC and Placebo: The tuberculosis subjects inject 1μg/ml ESAT6-CFP10 and the placebo of ESAT6-CFP10 only one time in the different time .Right arm inject ESAT6-CFP10 and left arm the placebo.Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml the placebo by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
- Tuberculosis Subjects- 5μg/ml EC and Placebo: The tuberculosis subjects inject 5μg/ml ESAT6-CFP10 and the placebo of ESAT6-CFP10 only one time in the different time .Right arm inject ESAT6-CFP10 and left arm the placebo.Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml the placebo by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
- Tuberculosis Subjects- 10μg/ml EC and Placebo: The tuberculosis subjects inject 10μg/ml ESAT6-CFP10 and the placebo of ESAT6-CFP10 only one time in the different time .Right arm inject ESAT6-CFP10 and left arm the placebo.Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml the placebo by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
- Tuberculosis Subjects- 20μg/ml EC and Placebo: The tuberculosis subjects inject 20μg/ml ESAT6-CFP10 and the placebo of ESAT6-CFP10 only one time in the different time .Right arm inject ESAT6-CFP10 and left arm the placebo.Two drugs must be use in the same subjects. Left arm intradermally inject with 0.1ml the placebo by a syringe(1ml).Observe 30 minutes , if without obvious adverse reaction then right arm intradermally inject with 0.1ml ESAT6-CFP10 by a syringe(1ml).
Arm/Group | Healthy Subjects-1μg/ml ECand TB-PPD | Healthy Subjects-5μg/ml EC and TB-PPD | Healthy Subjects-10μg/ml EC and TB-PPD | Healthy Subjects-20μg/ml EC and TB-PPD | Tuberculosis Subjects- 1μg/mlEC and TB-PPD | Tuberculosis Subjects- 5μg/ml EC and TB-PPD | Tuberculosis Subjects- 10μg/ml EC and TB-PPD | Tuberculosis Subjects- 20μg/ml EC and TB-PPD | Tuberculosis Subjects- 1μg/ml EC and Placebo | Tuberculosis Subjects- 5μg/ml EC and Placebo | Tuberculosis Subjects- 10μg/ml EC and Placebo | Tuberculosis Subjects- 20μg/ml EC and Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/14 | 6/14 | 1/14 | 1/14 | 4/14 | 4/14 | 2/14 | 3/14 | 0/8 | 3/8 | 4/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Subjects-1μg/ml ECand TB-PPD (N=14) | Healthy Subjects-5μg/ml EC and TB-PPD (N=14) | Healthy Subjects-10μg/ml EC and TB-PPD (N=14) | Healthy Subjects-20μg/ml EC and TB-PPD (N=14) | Tuberculosis Subjects- 1μg/mlEC and TB-PPD (N=14) | Tuberculosis Subjects- 5μg/ml EC and TB-PPD (N=14) | Tuberculosis Subjects- 10μg/ml EC and TB-PPD (N=14) | Tuberculosis Subjects- 20μg/ml EC and TB-PPD (N=14) | Tuberculosis Subjects- 1μg/ml EC and Placebo (N=8) | Tuberculosis Subjects- 5μg/ml EC and Placebo (N=8) | Tuberculosis Subjects- 10μg/ml EC and Placebo (N=8) | Tuberculosis Subjects- 20μg/ml EC and Placebo (N=8)
Itching at the injection site (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (3) | 1 (2) | 1 (1) | 3 (4) | 3 (5) | 1 (2) | 3 (5) | 0 (0) | 2 (2) | 3 (3) | 3 (3) — Itching at the injection site is the most common adverse events for this clinical trial .And the vast majority of itching is the first level(mild) .
Pain at the injection site (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
fever (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
High blood pressure (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Percentage abnormal of Eosinophils (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other